CLINICAL TRIAL: NCT01712646
Title: The Use of Daily, Intranasal Oxytocin for the Treatment of Childhood-Onset Schizophrenia (COS), a Randomized Double-Blind Trial
Brief Title: Daily Intranasal Oxytocin for Childhood-Onset Schizophrenia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 130004; 13-M-0004
Record Dates: First submitted 2012-10-20; First posted 2012-10-23 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2016-06-20

CONDITIONS: Childhood Onset Psychotic Disorders; Schizophrenia
Keywords: Oxytocin; Childhood Onset Schizophrenia; Double Blind
MeSH Terms: conditions — Schizophrenia; Schizophrenia, Childhood

INTERVENTIONS:
Drug: Intranasal Oxytocin

SUMMARY:
Background:

- Oxytocin is a chemical that the brain normally produces. It plays an important part in the way humans and other animals act in social and emotional situations. Adults with schizophrenia have been studied to see if oxytocin can reduce some symptoms of schizophrenia, such as hearing voices, feeling suspicious, and not feeling interested in daily life. These studies show that oxytocin may help. However, it has not been studied in children who develop schizophrenia. Researchers want to see if oxytocin, given as a nasal spray, is safe and can reduce schizophrenia symptoms in children.

Objectives:

- To see if an oxytocin nasal spray can reduce schizophrenia symptoms in children.

Eligibility:

- Children above 10 years of age who have childhood-onset schizophrenia, and have schizophrenia symptoms in spite of taking medication.

Design:

* This study will last 4 weeks. Participants will stay in the hospital for the entire period of the study. Participants may also have an extra 2 weeks of study medication and 1 week of testing immediately following the initial 4 weeks.
* Participants will be screened with a physical exam and medical and psychiatric history. They will provide blood and urine samples, and have imaging studies of the brain. They will also have tests to look at their social and emotional functioning. These tests will take 1 week to perform.
* Participants will have either oxytocin or placebo nasal spray twice daily for 2 weeks.
* At the end of the 2-week period with nasal spray, there will be 1 week with no nasal spray. All the tests of week 1 will be repeated.
* The optional extra 3 weeks (2 weeks with oxytocin and one week for testing) will be similar to the second, third, and fourth weeks of the study. All participants will have oxytocin during this period.

DETAILED DESCRIPTION:
Background:

Recent studies with intranasal oxytocin administration indicate moderate efficacy in symptom reduction in adult patients with schizophrenia, and moderate to good response in improving social cognition in patients with autism. The majority (about 75%) of patients with childhood-onset schizophrenia (COS) continue to show impairing social and psychotic symptoms after drug treatment optimization, and almost 30% of children with COS have co-morbid autism spectrum disorder (ASD). Oxytocin may be a safe and effective adjunctive treatment to improve social cognition, reduce anxiety, and indirectly reduce psychotic symptoms in medication-stable COS patients.

Objective:

To study whether intranasal oxytocin (study medication) would be safe, improve emotional/social cognition, and reduce symptom severity in clinically stable COS children and whether the study medication would also result in specific neurocircuitry changes, as measured by multimodal neuroimaging.

Study Population:

72 patients (36 per group) with COS, ages 10 and above will be recruited. All patients will be on stable medications for at least one month prior to this study.

Design:

Two-week double-blind, placebo-controlled, parallel design trial of daily intranasal oxytocin. Subsequent to the study period, a two-week extension of open label study medication will be offered to all participants, regardless of study group assignment.

Outcome Measures:

Primary Outcome Measures:

To evaluate the safety of intranasal oxytocin in COS patients.

To assess whether intranasal administration of oxytocin will improve both positive and negative symptoms of schizophrenia compared to placebo, as measured by PANSS, SAPS, SANS, and BPRS.

To evaluate whether intranasal oxytocin has significant effects on the social and emotional processing and behavior of children with COS, as measured by the Diagnostic Analysis of Nonverbal Behavior (DANVA-2), Developmental Neuropsychological Assessment (NEPSY-2) standardized social perception battery, Brune Theory of Mind Pictures Stories Task, Reading the Mind in the Eyes Test. Social Responsiveness Scale (SRS).

To measure alterations in neurocircuitry after oxytocin administration, as measured by fMRI, DTI, and MEG.

To evaluate changes in blood plasma oxytocin levels measured over the course of the study.

ELIGIBILITY:
* INCLUSION CRITERIA:

COS patients (age 10 and above) recruited, enrolled, and diagnosed under the screening protocol 03-M-0035.

Have been stable on their medications for at least one month prior to enrollment in this study, with the exception of occasional use of prn (as needed) medication. There are no contraindications to oxytocin; therefore, all medications are permitted.

Continued problems in social/emotional domains, as evidenced by problems with interpersonal relationships (e.g., poor ability to relate with others, make friends, have meaningful social interactions), emotional processing (e.g., difficulty interpreting emotions, inappropriate emotional responses, significant anxiety around activities of daily living, lack of empathy), and/or residual symptoms of schizophrenia (e.g., hallucinations, delusions, flat affect, disorganized thinking/behavior), despite medication.

EXCLUSION CRITERIA:

Any major neurological illness (e.g., epilepsy, brain tumors, metabolic disorders).

Is pregnant, plans on becoming pregnant during the study, or is actively breast-feeding.

Ages: 10 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-10-05; Primary Completion 2016-06-20 (Actual)

PRIMARY OUTCOMES:
Blood plasma oxytoxin levels
Neuocircuitry alterations in amygdale/cingulated
Brain activity alterations during exposure to social stimuli
Improved psychosis/anxiety symptoms
Improved DANVA-2/NEPSY-2/social interaction scores

CONTACTS AND LOCATIONS:
Overall Officials: Judith L Rapoport, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Asarnow JR, Ben-Meir S. Children with schizophrenia spectrum and depressive disorders: a comparative study of premorbid adjustment, onset pattern and severity of impairment. J Child Psychol Psychiatry. 1988 Jul;29(4):477-88. doi: 10.1111/j.1469-7610.1988.tb00738.x. PMID 3215919
- [Background] Watkins JM, Asarnow RF, Tanguay PE. Symptom development in childhood onset schizophrenia. J Child Psychol Psychiatry. 1988 Nov;29(6):865-78. doi: 10.1111/j.1469-7610.1988.tb00759.x. PMID 3235494
- [Background] Russell AT, Bott L, Sammons C. The phenomenology of schizophrenia occurring in childhood. J Am Acad Child Adolesc Psychiatry. 1989 May;28(3):399-407. doi: 10.1097/00004583-198905000-00017. PMID 2738007
- [Derived] Berman RA, Gotts SJ, McAdams HM, Greenstein D, Lalonde F, Clasen L, Watsky RE, Shora L, Ordonez AE, Raznahan A, Martin A, Gogtay N, Rapoport J. Disrupted sensorimotor and social-cognitive networks underlie symptoms in childhood-onset schizophrenia. Brain. 2016 Jan;139(Pt 1):276-91. doi: 10.1093/brain/awv306. Epub 2015 Oct 22. PMID 26493637